CLINICAL TRIAL: NCT04331275
Title: Viral Specific T-cells (VSTs) for Treatment of Viral Infections After Solid Organ Transplant
Brief Title: Viral Specific T-cells for Treatment of Viral Infections After Solid Organ Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoxworth Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0042
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Solid Organ Transplant; Viral Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viral Specific T-cells (VSTs) (Experimental)
  Interventions: Biological: Viral Specific T-cells (VSTs)

INTERVENTIONS:
Biological: Viral Specific T-cells (VSTs) — VSTs will be infused into solid organ transplant recipients who have evidence of viral infection.

SUMMARY:
The purpose of this research study is to learn more about the use of viral specific T-lymphocytes (VSTs) to treat viral infections that may happen after solid organ transplant (SOT). VSTs are cells specially designed to fight viral infections that may happen after a solid organ transplant. These cells are created from a blood sample collected from the study participant.

Solid organ transplant and the use of immunosuppressive medications reduces the body's ability to fight infections. Viral infections are a common problem after transplant and can cause significant complications. Reduction of immunosuppression may put the organ at risk of rejection. Moreover, treatment of viral infections is expensive and time consuming, with families often administering prolonged treatments with intravenous anti-viral medications, or patients requiring prolonged admissions to the hospital. The medicines can also have side effects like damage to the kidneys or reduction in the blood counts, so in this study the investigators are trying to find a better way to treat these infections and minimize complications.

ELIGIBILITY:
Inclusion Criteria:

* Blood adenovirus PCR ≥1,000
* Blood CMV PCR ≥ 500
* Blood EBV PCR ≥ 1,000
* Plasma BKV PCR >1,000
* Plasma JC Virus PCR > 1,000
* Evidence of invasive adenovirus infection. Adenovirus infection will be defined as the presence of adenoviral positivity as detected by PCR or culture from one site such as stool or blood or urine or nasopharynx. Adenovirus disease will be defined as the presence of adenoviral positivity as detected by culture or PCR from more than 2 sites such as stool or blood or urine or nasopharynx.
* Evidence of invasive CMV infection, e.g. pneumonitis, retinitis, colitis.
* Evidence of EBV-associated lymphoproliferation (EBV-LPD) defined as proven EBV-LPD by biopsy or probable EBV-LPD defined as an elevated EBV DNA level in the blood associated with clinical symptoms (adenopathy or fever or masses on imaging) but without biopsy confirmation.
* Evidence of symptomatic BK virus infection, which may include symptomatic hemorrhagic cystitis, BK viruria or BK nephropathy
* Evidence of PML or other CNS infection due to JC virus
* Clinical status must allow tapering of steroids to < 0.5mg/kg prednisone or other steroid equivalent, or a clinically acceptable steroid dose at the discretion of the PI
* Age > 1 day
* Must be able to receive VST infusion in Cincinnati

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Successful production of viral specific T-cells | Within 30 days post culture initiation
  Of the patients who had a VST culture initiated, successful production of VST cells is defined as meeting the protocol-defined release criteria.

SECONDARY OUTCOMES:
Presence of viral-specific T-cells | At 30 days after infusion
  Presence of viral-specific T-cells in the participant's blood will be assessed by Elispot assay

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States